CLINICAL TRIAL: NCT04169607
Title: Effect of Intraoperative Dynamic Compliance Guided Individualized Positive End-expiratory Pressure on Postoperative Atelectasis After Laparoscopic Bariatric Surgery: a Single-center, Double-blind Randomized Controlled Trial
Brief Title: Effect of Intraoperative Dynamic Compliance Guided Individualized Positive End-expiratory Pressure on Postoperative Atelectasis After Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XYFY2019-KL168-01
Record Dates: First submitted 2019-10-13; First posted 2019-11-20 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Atelectasis
Keywords: lung protective ventilation strategy; individualized positive end-expiratory pressure; Laparoscopic bariatric surgery; Mechanical ventilation; Anesthetic management; Lung dynamic compliance; Postoperative Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized PEEP (Experimental): Basic ventilation: Volume-controlled ventilation mode with positive end-expiratory pressure（PEEP） of 8cm H2O after induction of anesthesia，
  Recruitment maneuver: Pressure-controlled ventilation mode increasing PEEP from 10 to 25cmH2O.
  PEEP-titration maneuver: At this PEEP level, a decremental PEEP-titration maneuver will be started in volume-controlled ventilation mode, decreasing PEEP to 5cmH2O to confirm the highest dynamic lung compliance.
  After titration: A new recruitment maneuver will be performed and the final PEEP will be the one related to the highest dynamic lung compliance plus 2cm H2O.
  Randomization: Subsequently patient was randomized, the PEEP was then maintained (individualized PEEP arm) until extubation.
  After discharged from post-anesthesia care unit (60 to 90 minutes after extubation)：A chest computerized tomography（CT） will be performed to assess the amount of atelectasis, expressed as the percentage of lung tissue in CT.
  Interventions: Procedure: Dynamic compliance guided individualized positive end-expiratory pressure titration strategy
- PEEP 8 (Active Comparator): Bacis ventilation: Volume-controlled ventilation mode with positive end-expiratory pressure（PEEP） of 8cm H2O after induction of anesthesia，
  Recruitment maneuver: Pressure-controlled ventilation mode increasing PEEP from 10 to 25cmH2O.
  PEEP-titration maneuver: At this PEEP level, a decremental PEEP-titration maneuver will be started in volume-controlled ventilation mode, decreasing PEEP to 5cmH2O to confirm the highest dynamic lung compliance.
  After titration: A new recruitment maneuver will be performed and the final PEEP will be the one related to the highest dynamic lung compliance plus 2cm H2O.
  Randomization: Subsequently patient was randomized , the PEEP was then reduced to 8cm H2O (PEEP8 arm) until extubation.
  After discharged from post-anesthesia care unit (60 to 90 minutes after extubation)：A chest computerized tomography（CT） will be performed to assess the amount of atelectasis, expressed as the percentage of lung tissue in CT.
  Interventions: Procedure: Dynamic compliance guided individualized positive end-expiratory pressure titration strategy

INTERVENTIONS:
Procedure: Dynamic compliance guided individualized positive end-expiratory pressure titration strategy — Basic ventilation: Volume-controlled ventilation (VCV) mode with positive end-expiratory pressure (PEEP) of 8cm H2O after induction of anesthesia，
  Recruitment maneuver (RM): Pressure-controlled ventilation (PCV) mode increasing PEEP from 10 to 25cmH2O in step of 5cmH2O per 30s.
  PEEP-titration maneuver: ventilation parameters reset as basic ventilation with PEEP still 25cmH2O.Decrease PEEP to 5cmH2O in step of 2cmH2O per 10 respiratory cycles to confirm the highest dynamic lung compliance (Cdy).
  After titration: A new RM will be performed and the final PEEP will be the one related to highest Cdy plus 2cm H2O.
  Randomized after the second RM. Individualized PEEP arm: maintain individualized PEEP; PEEP8 arm: maintain a fixed PEEP of 8cm H2O.
  VCV with other ventilation parameters the same as basic ventilation until extubation .
  After discharged from postoperative anesthesia care unit (60 to 90 minutes after extubation): chest CT .

SUMMARY:
This study intends to explore the effect of dynamic compliance guided individualized positive end-expiratory pressure titration strategy on reducing the level of postoperative atelectasis in obese patient who have laparoscopic bariatric surgery.The results of the study are to assess the effects of this intervention on the incidence，duration of postoperative atelectasis and other complications including hypoxemia etc. after laparoscopic bariatric surgery.And reducing the burden of postoperative atelectasis on patients and their families, hospitals and public resources.

ELIGIBILITY:
Inclusion Criteria:

1. Bmi ≥ 35 kg/ m2
2. over 18 years old
3. elective laparoscopic bariatric surgery (gastric bypass or sleeve)

Exclusion Criteria:

1. ASA >IV
2. Lung bullae
3. thoracic surgery history
4. quit smoking less than 1 week
5. chronic obstructive pulmonary disease requiring oxygen
6. congestive heart failure (New York Heart Association classification ≥ III)
7. planned to be transferred to intensive care unit after surgery
8. Patients participating in another interventional study
9. Refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Percentage of postoperative atelectasis | 60-90 minutes after extubation
  The amount of postoperative atelectasis, expressed as the percentage of lung tissue in CT.

SECONDARY OUTCOMES:
pulse oxygen | 24 hours after surgery
  Continuous measurement of 24h pulse oxygen after surgery（%）
PaO2/FiO2 ratio | 1 day before surgery(baseline)，5 minutes after anesthesia induction，1 hour after pneumoperitoneum，before extubation，30 minutes after extubation
  PaO2/FiO2 ratio
Quality of Recovery Score - 40 (QoR-40) | 1 day before surgery(baseline)，1，2，7，30 days after surgery
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
Mini-Mental score examination (MMSE) | 1 day before surgery(baseline)，1，2 days after surgery
  Mini-Mental score examination [MMSE] used for screening of dementia.The total score on the MMSE ranges from 0 (most severe dementia) to 24 (no dementia).
Postoperative Complication | 1，2，7 days after surgery
  including pulmonary and other systematic postoperative complications
Mean arterial pressure | every 5minutes During Surgery；end of each step during RM and titration strategy
  Mean arterial pressure = (systolic blood pressure + 2 × diastolic blood pressure) / 3（mmHg）
systolic blood pressure | every 5minutes During Surgery；end of each step during RM and titration strategy
  systolic blood pressure measured by invasive arterial blood pressure（mmHg）
diastolic blood pressure | every 5minutes During Surgery；end of each step during RM and titration strategy
  diastolic blood pressure measured by invasive arterial blood pressure（mmHg）
heart rate | every 5minutes During Surgery；end of each step during RM and titration strategy
  heart rate per minute
pulse oxygen | every 5minutes During Surgery；end of each step during RM and titration strategy
  pulse oxygen（%）
dynamic compliance | every 5minutes During Surgery；end of each step during RM and titration strategy
  tidal volume/(airway peak pressure - PEEP)（ml/cmH2O）
airway plateau pressure | every 5minutes During Surgery；end of each step during RM and titration strategy
  airway plateau pressure is directly showed in the screen of ventilator（cmH2O）
airway peak pressure | every 5minutes During Surgery；end of each step during RM and titration strategy
  airway peak pressure is directly showed in the screen of ventilator（cmH2O）

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Li X, Liu H, Wang J, Ni ZL, Liu ZX, Jiao JL, Han Y, Cao JL. Individualized Positive End-expiratory Pressure on Postoperative Atelectasis in Patients with Obesity: A Randomized Controlled Clinical Trial. Anesthesiology. 2023 Sep 1;139(3):262-273. doi: 10.1097/ALN.0000000000004603. PMID 37440205